CLINICAL TRIAL: NCT00095537
Title: Phase I Study of BMS-599626 in Patients With Advanced Solid Malignancies, Including Malignancies That Express HER2 at the Maximum Tolerated Dose and/or Recommended Phase II Dose
Brief Title: BMS-599626 in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA181-002
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-10

CONDITIONS: Cancer; Metastases
Keywords: Solid tumors; cancer; HER-2-expressing tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — (4-((1-(3-fluorophenyl)methyl)-1H-indazol-5-ylamino)-5-methylpyrrolo(2,1-f)(1,2,4)triazin-6-yl)carbamic acid 3-morpholinylmethyl ester

ARMS (1):
- Phase 1 MTD Study (Experimental)
  Interventions: Drug: panHer

INTERVENTIONS:
Drug: panHer — Tablets, Oral, A modified Fibonocci dose escalation system initiated at 100mg and escalating up to 880mg maximum dose (rounded down to 20mg increments based on smallest tablet size); -2 40mg -33%; -1 60mg -40%; 1 100mg --; 2 200mg 100%; 3 320mg 67%; 4 480mg 50%; 5 660mg 40%; 6 880mg 33.3%, Daily, Until DLT or study MTD is reached.
  Other Names: BMS-599626

SUMMARY:
The purpose of this trial is to identify the highest oral dose of BMS-599626, a drug that is directed against EGFR and HER2 proteins, that can be given safely on a daily schedule of 21 days with a 7 day rest period in patients with cancer who no longer benefit from other commonly used treatments. The study will also test for other proteins that may be affected by BMS-599626; and the level of study drug in the blood will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic cancer that has progressed on currently available therapies;
* At least 3 month life expectancy;
* Primary cancer must be solid (non-hematologic);
* Adequate bone marrow, liver & kidney function;
* Negative pregnancy test.

Exclusion Criteria:

* Serious, uncontrolled medical disorder;
* Individuals not willing or able to use an acceptable method to avoid pregnancy for the entire study period and for at least 3 months after the study;
* Pregnant or breastfeeding women;
* Patients with known brain metastasis;
* Uncontrolled or significant cardiovascular disease;
* Anticancer therapy within 2-6 weeks prior to study drug (depending on the therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-03; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Det. the max tolerated dose,biologically active doses & recommended phase 2 dose of BMS-599626 when adm. as a daily oral dose to pts with HER2 expressing-metastatic solid tumors who have progressed on or following standard therapy

SECONDARY OUTCOMES:
Evaluate the effect of BMS-599626 on biomarkers & predictive markers of HER1/2 in skin metabolic act. through PET imaging & preliminary evidence of anti-tumor act.,determine the effect of gastric acid modifying agents on systemic exposure of BMS-599626

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Los Angeles, California